CLINICAL TRIAL: NCT04327336
Title: Effectiveness of Noninvasive Ventilation Adjusted Automatically in the Obesity Hypoventilation Syndrome
Brief Title: Randomized Controlled Trial Between Auto-titration and Manual Titration of Non-invasive Ventilation in Obesity Hypoventilation Syndrome
Acronym: TITRATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Juan F. Masa, Principal Investigator, Sociedad Española de Neumología y Cirugía Torácica
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI16/01704
Record Dates: First submitted 2018-05-15; First posted 2020-03-31 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Chronic Hypercapnic Respiratory Failure; Obesity Hypoventilation Syndrome
Keywords: Chronic respiratory failure; Obesity; Non invasive mechanical ventilation
MeSH Terms: conditions — Obesity Hypoventilation Syndrome; Obesity

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, double arm, double blind controlled trial.
Who Masked: Participant, Investigator
Masking Description: Two investigators (named Investigator 1 and Investigator 2) participate in each center, with different tasks. Investigator 1 is responsible of randomization and will be aware of the study group assigned to the patient. Investigator 2 will collect in each visit health resource utilization, specific and QoL tests and laboratory test results. Investigator 2 does not know the study arm.
  Patients will not be informed about the ventilator settings and the menu of the ventilator will be locked, so they cannot access to ventilator data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual (Active Comparator): In this group non invasive mechanical ventilation will be manually titrated during a polysomnography. The Philips A40 ventilator will be used in Spontaneous-Timed (ST) mode.
  Interventions: Device: Manual Non invasive ventilation titration
- Automatic (Active Comparator): In this group the ventilator will run in an automatic mode (AVAPS) with the same Phillips A40 ventilator.
  Interventions: Device: Automatic Non invasive ventilation titration

INTERVENTIONS:
Device: Manual Non invasive ventilation titration — Manual Group: during a complete polysomnography, adding transcutaneous capnography and the basic ventilators curves, the ventilators setting will be adjusted in order to correct respiratory events and patient-ventilator asyncrony. A 10 hours face-to-face investigator training meeting is programmed before opening the inclusion period.
  Arms: Manual
Device: Automatic Non invasive ventilation titration — Automatic Group: the A40 ventilator in the automatic AVAPS mode will be adjusted in order to achieve 8-10 ml/kg of ideal weight.
  Arms: Automatic

SUMMARY:
Primary Objectives: To evaluate the effectiveness in the obesity hypoventilation syndrome (OHS) treatment with non-invasive ventilation (NIV) set manually by polysomnography compared to the same treatment with a respirator with automatic NIV adjustment, analyzing as primary variable PaCO2 and as operational variables dropout rate for medical reasons and mortality. Secondary objectives: cost-effectiveness, clinical and functional improvement in wakefulness and during sleep, quality of life, blood pressure monitoring for 24 hours, incidence and evolution of cardiovascular events and use of health resources. Other objectives: 1) effectiveness of treatments in the following subgroups of patients: gender, age, socioeconomic status, severity of sleep apnea, VNI compliance, quality of life and comorbidities; 2) To evaluate the profile of patients with poor adherence to NIV based on clinical severity, gender, age and socioeconomic status in the whole sample and in both intervention groups.

DETAILED DESCRIPTION:
Method: Prospective, blind researchers, randomized, controlled non-inferiority and cost-effectiveness relationship, with two parallel open groups. 200 OHS patients will be divided into two groups by simple randomization 1:1 and followed for one year. The premise of non-inferiority is -2 at the lower limit of the confidence interval 95% for the change in PCO2 between the arms being assessed by analysis of covariance, adjusted for 2-sided, age, sex, body mass index in intention-to-treat and per-protocol analysis. The cost-effectiveness will be performed by Bayesian techniques with sensitivity analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Obesity Hypoventilation Syndrome defined by obesity (IMC≥30) and Hypercapnic respiratory failure (PCO 2> 45 mm Hg) in stable phase (PH≥7.35 without clinical signs of worsening in at least one previous month).
2. Age between 18-80 years.
3. Absence of other diseases causing hypercapnia as moderate or severe chronic obstructive pulmonary disease (FEV1> 70% predicted if FEV1 / FVC <70), neuromuscular, thoracic wall or metabolic disease; d) Absence of narcolepsy or restless legs syndrome.
4. Overcome correctly a 30 minutes test of treatment with VNI in wakefulness.

Exclusion Criteria:

1. Psychophysical disability for questionnaires.
2. Patients who cannot be evaluated by quality of life questionnaires because they present debilitating chronic disease.
3. Chronic nasal obstruction that prevents the use of NIV.
4. Pregnancy.
5. No informed consent obtained.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Change in PaCO2 between arms | 1 year
  Arterial blood gases while room air breathing expressed in mmHg

SECONDARY OUTCOMES:
Cost-effectiveness analysis by primary outcome | 1 year
  Cost-effectiveness analysis based on the primary outcome in mmHg Differences in within trial costs will be related with the differences in effectiveness (primary outcome) between arms using a probabilistic Bayesian approach to calculate the cost-effectiveness plane.
Cost-effectiveness analysis by QALY | 1 year
  Cost-effectiveness analysis based on the quality adjusted life year (QALY) Differences in within trial costs will be related with the differences in effectiveness (QALY) between arms using a probabilistic Bayesian approach to calculate the cost-effectiveness plane.
Change in subjective daytime sleepiness | 1 year
  Sleepiness evaluated by Epworth sleepiness scale, range from 0 to 24, being 0 the best result and 24 the worst.
Change in Quality of life measured by Functional Sleep Outcomes of Sleep Questionnaire (FOSQ) | 1 year
  Quality of life measured by Functional Sleep Outcomes of Sleep Questionnaire (FOSQ), range from 0 to 120, being 0 the worst result and 120 the best result .
Change in Quality of life measured by visual analogical wellbeing scale (VAWS) | 1 year
  Quality of life measured by visual analogical well-being scale (VAWS), range from 0 to 100, being 0 the worst result and 120 the best result .
Change in Quality of life measured by Euroqol 5D. | 1 year
  Quality of life measured by Euroqol 5D, range from 0 to 1, being 0 the worst result and 1 the best result .
Change in Quality of life measured by Short Form-36 (SF36), Mental component | 1 year
  Quality of life measured by Short Form-36 (SF36) Mental component,range from 0 to 100, being 0 the worst result and 100 the best result.
Change in Quality of life measured by Short Form-36 (SF36), Physical component | 1 year
  Quality of life measured by Short Form-36 (SF36) Physical component,range from 0 to 100, being 0 the worst result and 100 the best result.
Change in Bicarbonate arterial blood concentration | 1 year
  Arterial blood gases while breathing room air expressed in mmol/L
Change in PaO2 | 1 year
  Arterial blood gases while breathing room air expressed PaO2 in mmHg
Change in pH | 1 year
  Arterial blood gases while breathing room air
Change in polysomnographic Sleep periods | 1 year
  Standard polysomnography. time of sleep periods (Stage 1,2,3,4 and REM) in minutes.
Change in Arousal Index | 1 year
  Standard polysomnography, number of arousals per sleep hour
Change in Apnea-Hypopnea index | 1 year
  Standard polysomnography, number of apneas and hypoapneas per sleep hour
Change in Oxygen desaturation index | 1 year
  Standard polysomnography, number of 3% or more Oxygen desaturations per sleep hour
Change in Sleep time with Oxygen saturation below 90% | 1 year
  Standard polysomnography, percentage of sleep time with oxygen saturation below 90%
Change in polysomnographic parameters: Total Sleep time (TTS) | 1 year
  Standard polysomnography, time in minutes
Change in the blood pressure monitoring | at baseline and after a year
  The blood pressure will be monitored during 24 hours with a Blood Pressure Monitoring device before (baseline) and after intervention (1 year) in both arms measured in mmHg. Change in the mean blood pressure will be compared between arms
Incidental cardiovascular events | 1 year
  New hypertension diagnosis or anti-hypertensive treatment, atrial fibrillation, hospitalization for nonfatal myocardial infarction or instable angina, nonfatal stroke or transient ischemic attack or for heart failure episode, and cardiovascular death. Data obtained from official electronic health care databases
Health care resources utilization: Hospital admission | 1 year
  Hospital admission measured in number of events
Health care resources utilization: Hospital duration | 1 year
  Hospital duration measured in days of hospitalization
Health care resources utilization: ICU admission | 1 year
  ICU admission measured in numbers of events
Health care resources utilization: ICU duration | 1 year
  ICU duration measured in days of UCI admissions
Health care resources utilization: emergency visits | 1 year
  Emergency visits measured in number of events
Health care resources utilization: primary care visits | 1 year
  Primary care visits measured in number of events
Health care resources utilization: specialist visits | 1 year
  Specialist visits measured in number of events
Incidence of new adverse event | 1 year
  Number of adverse events based in CTCAE v4.0
Side effects | 1 year
  Incidence or side effects of NIV in follow-up visits: excessive noise, headache, claustrophobia, difficulty in sleep conciliation or maintenance, expiration discomfort.

OTHER OUTCOMES:
Adherent vs. non-adherent to noninvasive ventilation therapy subgroups | 1 year
  Efficacy between arms measuring Epworth sleepiness scale (from 0 to 24 points) comparing adherent vs. non-adherent to non-invasive ventilation therapy subgroups (higher and lower of 4 hours per day)
Sleep apnea severity subgroup | 1 year
  Efficacy between arms measuring Epworth sleepiness scale (from 0 to 24 points) comparing sleep apnea severity subgroups measured by apnea and hypopnea index at baseline (higher and lower of the median)
Hypercapnia severity subgroup | 1 year
  Efficacy between arms measuring Epworth sleepiness scale (from 0 to 24 points) comparing hypercapnia severity subgroups measured by PaCO2 (mmHg) at baseline (higher and lower of the median)
Systemic hypertension subgroup | 1 year
  Efficacy between arms measuring Epworth sleepiness scale (from 0 to 24 points) comparing the presence of hypertension diagnosis subgroups at baseline
Hypercapnia resolution subgroup | 1 year
  Efficacy between arms measuring Epworth sleepiness scale (from 0 to 24 points) comparing the resolution of hypercapnia measured by PaCO2 (mmHg) at the end of the follow-up (higher and lower of 45 mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Juan F Masa, PhD, Principal Investigator — Hospital San Pedro de Alcantara
Locations (1):
- Juan F. Masa, Cáceres, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mokhlesi B, Kryger MH, Grunstein RR. Assessment and management of patients with obesity hypoventilation syndrome. Proc Am Thorac Soc. 2008 Feb 15;5(2):218-25. doi: 10.1513/pats.200708-122MG. PMID 18250215
- [Background] Nowbar S, Burkart KM, Gonzales R, Fedorowicz A, Gozansky WS, Gaudio JC, Taylor MR, Zwillich CW. Obesity-associated hypoventilation in hospitalized patients: prevalence, effects, and outcome. Am J Med. 2004 Jan 1;116(1):1-7. doi: 10.1016/j.amjmed.2003.08.022. PMID 14706658
- [Background] Berg G, Delaive K, Manfreda J, Walld R, Kryger MH. The use of health-care resources in obesity-hypoventilation syndrome. Chest. 2001 Aug;120(2):377-83. doi: 10.1378/chest.120.2.377. PMID 11502632
- [Background] Lopez-Jimenez MJ, Masa JF, Corral J, Teran J, Ordaz E, Troncoso MF, Gonzalez-Mangado N, Gonzalez M, Lopez-Martinez S, De Lucas P, Marin JM, Marti S, Diaz-Cambriles T, Diaz-de-Atauri J, Chiner E, Aizpuru F, Egea C, Romero A, Benitez JM, Sanchez-Gomez J, Golpe R, Santiago-Recuerda A, Gomez S, Barbe F, Bengoa M; Grupo cooperativo. Mid- and Long-Term Efficacy of Non-Invasive Ventilation in Obesity Hypoventilation Syndrome: The Pickwick's Study. Arch Bronconeumol. 2016 Mar;52(3):158-65. doi: 10.1016/j.arbres.2015.10.003. Epub 2015 Dec 4. English, Spanish. PMID 26656679
- [Background] Masa JF, Celli BR, Riesco JA, Hernandez M, Sanchez De Cos J, Disdier C. The obesity hypoventilation syndrome can be treated with noninvasive mechanical ventilation. Chest. 2001 Apr;119(4):1102-7. doi: 10.1378/chest.119.4.1102. PMID 11296176
- [Background] Perez de Llano LA, Golpe R, Ortiz Piquer M, Veres Racamonde A, Vazquez Caruncho M, Caballero Muinelos O, Alvarez Carro C. Short-term and long-term effects of nasal intermittent positive pressure ventilation in patients with obesity-hypoventilation syndrome. Chest. 2005 Aug;128(2):587-94. doi: 10.1378/chest.128.2.587. PMID 16100142
- [Background] Janssens JP, Derivaz S, Breitenstein E, De Muralt B, Fitting JW, Chevrolet JC, Rochat T. Changing patterns in long-term noninvasive ventilation: a 7-year prospective study in the Geneva Lake area. Chest. 2003 Jan;123(1):67-79. doi: 10.1378/chest.123.1.67. PMID 12527605
- [Background] Masa JF, Corral J, Alonso ML, Ordax E, Troncoso MF, Gonzalez M, Lopez-Martinez S, Marin JM, Marti S, Diaz-Cambriles T, Chiner E, Aizpuru F, Egea C; Spanish Sleep Network. Efficacy of Different Treatment Alternatives for Obesity Hypoventilation Syndrome. Pickwick Study. Am J Respir Crit Care Med. 2015 Jul 1;192(1):86-95. doi: 10.1164/rccm.201410-1900OC. PMID 25915102
- [Background] Piper AJ, Wang D, Yee BJ, Barnes DJ, Grunstein RR. Randomised trial of CPAP vs bilevel support in the treatment of obesity hypoventilation syndrome without severe nocturnal desaturation. Thorax. 2008 May;63(5):395-401. doi: 10.1136/thx.2007.081315. Epub 2008 Jan 18. PMID 18203817
- [Background] Borel JC, Tamisier R, Gonzalez-Bermejo J, Baguet JP, Monneret D, Arnol N, Roux-Lombard P, Wuyam B, Levy P, Pepin JL. Noninvasive ventilation in mild obesity hypoventilation syndrome: a randomized controlled trial. Chest. 2012 Mar;141(3):692-702. doi: 10.1378/chest.10-2531. Epub 2011 Sep 1. PMID 21885724
- [Background] Berry RB, Chediak A, Brown LK, Finder J, Gozal D, Iber C, Kushida CA, Morgenthaler T, Rowley JA, Davidson-Ward SL; NPPV Titration Task Force of the American Academy of Sleep Medicine. Best clinical practices for the sleep center adjustment of noninvasive positive pressure ventilation (NPPV) in stable chronic alveolar hypoventilation syndromes. J Clin Sleep Med. 2010 Oct 15;6(5):491-509. PMID 20957853
- [Background] Gonzalez-Bermejo J, Perrin C, Janssens JP, Pepin JL, Mroue G, Leger P, Langevin B, Rouault S, Rabec C, Rodenstein D; SomnoNIV Group. Proposal for a systematic analysis of polygraphy or polysomnography for identifying and scoring abnormal events occurring during non-invasive ventilation. Thorax. 2012 Jun;67(6):546-52. doi: 10.1136/thx.2010.142653. Epub 2010 Oct 22. PMID 20971982
- [Background] Johnson KG, Johnson DC. Treatment of sleep-disordered breathing with positive airway pressure devices: technology update. Med Devices (Auckl). 2015 Oct 23;8:425-37. doi: 10.2147/MDER.S70062. eCollection 2015. PMID 26604837
- [Background] Jaye J, Chatwin M, Dayer M, Morrell MJ, Simonds AK. Autotitrating versus standard noninvasive ventilation: a randomised crossover trial. Eur Respir J. 2009 Mar;33(3):566-71. doi: 10.1183/09031936.00065008. PMID 19251798